CLINICAL TRIAL: NCT00174330
Title: A Multi-Center, Randomized, Open-Label Study To Evaluate Efficacy And Safety Of Dual Therapy With Atorvastatin Plus Amlodipine When Compared Amlodipine Therapy Alone In The Treatment Of Subjects With Concurrent Hyperlipidemia And Hypertension.
Brief Title: Comparing Amlodipine/Atorvastatin Co-Administration To Amlodipine Alone In Patients With Hypertension And Dyslipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3841026
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Atorvastatin; Amlodipine

INTERVENTIONS:
Drug: atorvastatin
Drug: amlodipine

SUMMARY:
To evaluate efficacy of the dual therapy of atorvastatin + amlodipine vs. amlodipine alone .

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of both hyperlipidemia and hypertension.

Exclusion Criteria:

* Subjects with Type 1 diabetes mellitus or Type 2 diabetes mellitus.
* Subjects with other atherosclerotic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330
Dates: Start 2005-05; Study Completion 2006-02

PRIMARY OUTCOMES:
To evaluate efficacy of the dual therapy of atorvastatin 10mg or 20mg + amlodipine 5mg or 10mg vs. amlodipine 5mg or 10mg alone

SECONDARY OUTCOMES:
To provide comparative evaluation of the safety profile of the dual therapy with atorvastatin + amlodipine versus amlodipine alone.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- China (9):
  - Pfizer Investigational Site, Beijing, Beijing Municipality
  - Pfizer Investigational Site, Guangzhou, Guangdong
  - Pfizer Investigational Site, Nanjing, Jiangsu
  - Pfizer Investigational Site, Shenyang, Liaoning
  - Pfizer Investigational Site, Shanghai, Shanghai Municipality
  - Pfizer Investigational Site, Hangzhou, Zhejiang
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Shanghai
  - Pfizer Investigational Site, Tianjin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3841026&StudyName=Comparing+Amlodipine%2FAtorvastatin+Co%2DAdministration+To+Amlodipine+Alone+In+Patients+With++Hypertension+And+Dyslipidemia+